CLINICAL TRIAL: NCT03655236
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of K0706 in Subjects With Early Parkinson's Disease
Brief Title: PROSEEK: A Phase 2 Study In Early Parkinson's Disease Patients Evaluating The Safety And Efficacy Of Abl Tyrosine Kinase Inhibition Using K0706
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated based on study outcomes
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_18_06
Record Dates: First submitted 2018-08-18; First posted 2018-08-31 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Early Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- K0706, low dose (Experimental)
  Interventions: Drug: K0706
- K0706, high dose (Experimental)
  Interventions: Drug: K0706
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: K0706 — low dose, orally, once-daily
  Arms: K0706, low dose
Drug: K0706 — high dose, orally, once-daily
  Arms: K0706, high dose
Other: placebo — placebo, orally, once-daily
  Arms: Placebo

SUMMARY:
This study consists of 2 parts. Part 1 of the study is conducted to evaluate the efficacy, safety, and tolerability of two doses of K0706 compared to placebo in subjects with early Parkinson's Disease who are not receiving dopaminergic therapy. Part 2 is an optional long term extension study for subjects who have completed week 40 of Part 1

DETAILED DESCRIPTION:
This study is designed to assess the ability of K0706 to slow the progression of PD. Preclinical animal model data have already demonstrated that K0706 has neuroprotective activity, but further development will require human clinical experience.

This study will also allow determination of safety and tolerability of K0706 over many months in subjects with PD.

ELIGIBILITY:
Part 1:

Inclusion criteria:

1. Males or females aged ≥ 50 years;
2. Body mass index (BMI) greater than 18.5 kg/m2 and less than 45 kg/m2;
3. Diagnosed with "Clinically Probable PD" according to the MDS clinical diagnostic criteria, with documented diagnosis of PD per treating physician's records within three years of the Screening visit. Disease severity according to modified Hoehn & Yahr stage ≤ 2;
4. Projected to not required to start dopaminergic therapy within 9 months from Baseline;

Exclusion criteria:

1. Current, or within 60 days of Screening, use of any prescription, investigational, or over the counter medication for the symptomatic treatment of PD or to slow the progression of PD. Treatment with Monoamine Oxidase B (MAOB) inhibitors will be allowed if the dose is stable for at least 30 days prior to Screening and subjects agree to remain on it for the duration of the study;
2. Prior use of dopaminergic therapy (e.g., levodopa, dopamine agonist, amantadine) for 30 or more days any time in the past;
3. A diagnosis of a significant central or peripheral nervous system disease affecting the subject's cognition or motor function at any time, such as another neurodegenerative disorder, multiple sclerosis or stroke. This does not include transient neurological deficits such as transient ischemic attacks or migraine aura;
4. A diagnosis of a medical condition that could interfere with interpretation of the MDS-UPDRS during the trial (e.g., musculoskeletal disorders);
5. Contraindications to receiving an MRI;
6. Contraindications to receiving a DaT SPECT scan (e.g., hypersensitivity to the active substance, any of the excipients, or iodine) if a new DaT SPECT scan is required for the study;
7. Most recent DaT SPECT scan not compatible with PD (i.e., Scans Without Evidence of Dopaminergic Deficit [SWEDD]) based on a central reading by a study physician;
8. MRI of the brain performed after onset of PD suggestive of secondary Parkinsonism (e.g., subdural hematoma, normal pressure hydrocephalus, or infarcts of the basal ganglia);
9. Severe tremors as defined by a score of "severe" on any of the MDS-UPDRS Parts 2 or 3 tremor severity (not constancy) items;
10. Montreal cognitive assessment score < 25
11. History of any surgery on the brain itself including deep brain stimulation for PD (note this does not include surgeries on the skull that do not affect the brain, e.g., small meningioma removal);
12. History of hypersensitivity (e.g., bronchospasm, anaphylaxis, serious drug rash) to contents of the study drug or other tyrosine kinase inhibitors;
13. Recent use of medications that can cause Parkinsonism and suspicion of the investigator that it could have worsened the subject's Parkinsonism. This includes neuroleptics (e.g., olanzapine, risperidone, haloperidol), some anti-nausea medications (e.g., prochlorperazine, metoclopramide) and others (e.g., flunarizine, methyldopa)
14. Use of medications that affect the dopaminergic system within 60 days of Screening. This includes stimulants (e.g., methylphenidate, amphetamine derivatives, modafinil) and Monoamine Oxidase A (MAOA) inhibitors (e.g., phenelzine, and tranylcypromine). Note that antidepressants are acceptable as long as the subject has remained on them at a stable dose for over 60 days prior to Screening and plans to remain on them through the study;
15. Any malignant disease (other than basal cell carcinoma of the skin) with evidence of disease within the past 5 years and with the potential for recurrence

Part 2:

Inclusion criteria:

1. Subject has completed part 1 of the study.
2. Subject projected not to need dopaminergic treatment except for treatment with Monoamine Oxidase B (MAOB) inhibitors. MAOB inhibitors will be allowed if the patient was already taking the same during part 1 of the study.
3. Subject has received K0706/placebo, as appropriate, within 4 weeks prior to end of part 1 of the study.
4. Male subjects enrolled in the study should not father a child and are advised to prevent the passage of semen to their sexual partner during intercourse using an effective method, as judged by the Investigator, for the duration of the study and for 3 months after the last dose of study drug

Exclusion criteria:

1. Clinically significant or unstable psychiatric or medical condition, vital sign, or laboratory abnormality that in the opinion of the investigator interferes with participation in the study
2. Any condition that in the opinion of the Investigator represents an obstacle for study conduct and/or represents a potential unacceptable risk for the subject.
3. Subject has any concurrent medical condition or uncontrolled, clinically significant systemic disease (e.g., renal failure, heart failure, hypertension, liver disease, diabetes, or anemia) that, in the opinion of the Investigator, could cause continued treatment to be detrimental to the subject

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (34):
  - Xenoscience Inc. - 21st Century Neurology, Phoenix, Arizona
  - University of Arkansas for Medical Sciences (UAMS) - Movement Disorders Clinic, Little Rock, Arkansas
  - Keck Hospital of USC, Los Angeles, California
  - Pacific Movement Disorders Center Pacific Neuroscience Institute Providence Saint John's Health Center, Santa Monica, California
  - Georgetown University Medical Center Department of Neurology, 7PHC, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Inc., Boca Raton, Florida
  - Neurology Associates PA, Maitland, Florida
  - Visionary Investigators Network, Miami, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Struthers Parkinson's Center -Park Nicollet, Golden Valley, Minnesota
  - Washington University (WUSTL) School of Medicine, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center (DHMC) Neurology Research, Lebanon, New Hampshire
  - Robert Wood Johnson Medical School Department of Neurology, Clinical Academic Building (CAB), New Brunswick, New Jersey
  - Neurology Specialists of Monmouth County, PA, West Long Branch, New Jersey
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Weill Cornell Medicine Department of Neurology Parkinson's Disease and Movement Disorders Institute, New York, New York
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Advanced Neurology Epilepsy and Sleep Center, El Paso, Texas
  - Baylor College of Medicine (BCM)- Parkinson's Disease Center and Movement Disorders Clinic (PDCMDC), Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Central Texas Neurology Consultants (CTNC), Round Rock, Texas
  - Evergreen Health, Kirkland, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Hungary (4):
  - Nyiro Gyula Hospital, Budapest, Buapest
  - Valeomed Diagnosztikai Kozpont, Esztergom, Komárom-Esztergom
  - Szent Borbála Kórház, Tatabánya, Komárom-Esztergom
  - Pest Megyei Flór Ferenc Kórház, Kistarcsa, Pest County
- India (12):
  - Nizam's Institute of Medical Sciences, Panjagutta, Hyderabad
  - P.D. Hinduja National Hospital and Medical Care Research Centre, Mumbai, Maharashtra
  - Jaslok Hospital and Research centre, Mumbai, Maharashtra
  - Fortis Flt. Lt. Rajan Dhall Hospital, Vasant Kunj, New Delhi
  - Medipoint Hospital, Aundh, Pune
  - Lifepoint Multispeciality Hospital Pvt Ltd, Wakad, Pune
  - Dayanand Medical College & Hospital, Research & Development Centre, Ludhiana, Punjab
  - Citi Neuro Centre, Hyderabad, Telangana
  - Institute of Neurosciences Kolkata, Kolkata, West Bengal
  - Bangur Institute of Neurosciences & Psychiatry (BINP), Kolkata
  - Sir Ganga Ram Hospital, New Delhi
  - Deenanath Mangeshkar Hospital & Research Center (DMHRC), Pune
- Poland (11):
  - NZOZ Centrum Medyczne HCP, Poznan, Greater Poland Voivodeship
  - Nasz Lekarz Przychodnie Medyczne Ośrodek Badań Klinicznych, Torun, Kuyavian-Pomeranian Voivodeship
  - Krakowska Akademia Neurologii, Krakow, Lesser Poland Voivodeship
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin, Lublin Voivodeship
  - ETG Lublin, Lublin, Lublin Voivodeship
  - RCMed Oddział w Sochaczewie, Sochaczew, Masovian Voivodeship
  - SINGUA Sp. Z o.o., Warsaw, Masovian Voivodeship
  - C.M. Silmedic Sp. z o.o., Katowice, Silesian Voivodeship
  - Neuro-Care - Sp. z o.o. Sp. Komandytowa Ul. Szpitalna 6, Siemianowice Śląskie, Silesian Voivodeship
  - Mazowiecki Szpital Brodnowski w Warszawie Sp. z o.o., Warsaw
  - SOMED CR, Lodz, Łódź Voivodeship
- Slovakia (3):
  - NEURES, s.r.o., Krompachy, Spiska Nova Ves
  - Medical Center Konzilium, Dubnica nad Váhom, Trenčín Region
  - MUDr. Beata Dupejova, neurologicka ambulancia s.r.o, Banská Bystrica
- Spain (14):
  - Plaza de Cruces, S/N, Barakaldo, Bilbao
  - Policlínica Gipuzkoa, Donostia / San Sebastian, San Sebastián
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari General de Catalunya, Barcelona
  - Hospital Universitari de Bellvitge (IDIBELL), Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Quiron Salud, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102

RESULTS

PARTICIPANT FLOW:
Groups:
- K0706, Low Dose: K0706: low dose, orally, once-daily. This study consists of two parts. Subjects received K0706, Low dose in Part 1 and Part 2 of the study. All subjects will continue treatment for up to 36 weeks
- K0706, High Dose: K0706: high dose, orally, once-daily This study consists of two parts. Subjects received K0706, high dose in Part 1 and Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
- Placebo: placebo: placebo, orally, once-daily This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. All subjects will continue treatment for up to 36 weeks.
Period: Subject Disposition in Part 1 Period
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Started | 171 | 174 | 168
Completed | 114 | 66 | 120
Not Completed | 57 | 108 | 48
Not completed — Adverse Event | 25 | 55 | 12
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Parkinson's disease progression | 2 | 8 | 5
Not completed — Poor compliance | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Requires prohibited medication | 4 | 5 | 3
Not completed — Study terminated by Sponsor | 12 | 8 | 13
Not completed — Withdrawal by Subject | 0 | 5 | 3
Not completed — Withdrawal of consent | 11 | 16 | 6
Not completed — Other | 0 | 2 | 2
Period: Subject Disposition in Part 2 Period
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Started | 72 | 40 | 77 (Prior placebo transitioned to K0706 high-dose)
Completed | 36 | 21 | 27
Not Completed | 36 | 19 | 50
Not completed — Adverse Event | 2 | 5 | 12
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Parkinson's disease progression | 4 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 4
Not completed — Requires prohibited medication | 3 | 1 | 5
Not completed — Study terminated by Sponsor | 18 | 11 | 13
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Withdrawal of consent | 5 | 1 | 12
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- K0706, Low Dose: K0706: low dose, orally, once-daily This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. Subjects that had been randomized to either dose of K0706 in part 1 of the study will continue on the same dosing regimen in Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
- K0706, High Dose: K0706: high dose, orally, once-daily This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. Subjects that had been randomized to either dose of K0706 in part 1 of the study will continue on the same dosing regimen in Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
- Placebo: placebo: placebo, orally, once-daily (Prior placebo transitioned to K0706 high-dose) This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. Subjects that had been randomized to either dose of K0706 in part 1 of the study will continue on the same dosing regimen in Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
- Total: Total of all reporting groups
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo | Total
Number analyzed (Participants) | 171 | 174 | 168 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Prior placebo transitioned to K0706 high-dose
  years
    Part 1 | 64.3 (8.44) | 65.3 (7.67) | 65.4 (8.03) | 65.0 (8.05)
    Part 2: number analyzed (Participants) | 72 | 40 | 77 | 189
    Part 2 | 62.6 (7.75) | 65.3 (6.66) | 66.0 (7.84) | 64.5 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Prior placebo transitioned to K0706 high-dose
  Participants
    Part 1: Female | 61 | 71 | 47 | 179
    Part 1: Male | 110 | 103 | 121 | 334
    Part 2: number analyzed (Participants) | 72 | 40 | 77 | 189
    Part 2: Female | 23 | 11 | 20 | 54
    Part 2: Male | 49 | 29 | 57 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Prior placebo transitioned to K0706 high-dose
  Participants
    Part 1: Hispanic or Latino | 16 | 17 | 15 | 48
    Part 1: Not Hispanic or Latino | 154 | 156 | 153 | 463
    Part 1: Unknown or Not Reported | 1 | 1 | 0 | 2
    Part 2: number analyzed (Participants) | 72 | 40 | 77 | 189
    Part 2: Hispanic or Latino | 8 | 2 | 4 | 14
    Part 2: Not Hispanic or Latino | 64 | 38 | 73 | 175
    Part 2: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Prior placebo transitioned to K0706 high-dose
  Participants
    Part 1: American Indian or Alaska Native | 0 | 0 | 1 | 1
    Part 1: Asian | 33 | 29 | 28 | 90
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Part 1: Black or African American | 6 | 1 | 3 | 10
    Part 1: White | 132 | 144 | 136 | 412
    Part 1: More than one race | 0 | 0 | 0 | 0
    Part 1: Unknown or Not Reported | 0 | 0 | 0 | 0
    Part 2: number analyzed (Participants) | 72 | 40 | 77 | 189
    Part 2: American Indian or Alaska Native | 0 | 0 | 1 | 1
    Part 2: Asian | 19 | 6 | 13 | 38
    Part 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Part 2: Black or African American | 1 | 1 | 0 | 2
    Part 2: White | 52 | 33 | 63 | 148
    Part 2: More than one race | 0 | 0 | 0 | 0
    Part 2: Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 40 in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Total Score.
Description: Part III: Motor examination: 18 items. Score range: 0-132, 32 and below is mild, 59 and above is severe.
Time Frame: Week 40
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
score on a scale | 1.5 (8.77) | 1 (7.58) | -1 (8.13)

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Time Frame: Part 2 (Week 40 to 80)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- K0706, Low Dose: K0706: low dose, orally, once-daily Subjects received K0706, Low dose in Part 1 and Part 2 of the study.
- K0706, High Dose: K0706: high dose, orally, once-daily Subjects received K0706, high dose in Part 1 and Part 2 of the study. In addition, subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40.
- Placebo: placebo: placebo, orally, once-daily Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40.
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 72 | 40 | 77
Participants | 37 | 24 | 61

3. Secondary Outcome: Part 1: Change From Baseline to Week 40 in the Sum of the MDS-UPDRS Part II and Part III Total Scores and Part 2: Change From Week 40 to Week 76 in the MDS-UPDRS Part III Total Score.
Description: The Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II assesses the motor aspects of experiences of daily living based on patient self-report. It comprises 13 items, each rated on a 5-point scale ranging from 0 (normal) to 4 (severe impairment). The total score for Part II ranges from 0 to 52, calculated as the sum of the individual item scores.
  The MDS-UPDRS Part III assesses the motor symptoms of Parkinson's disease. This part consists of 18 items, which are assessed across various body regions, resulting in 33 individual scores. Each item is rated on a 5-point scale from 0 (normal) to 4 (severe impairment), with higher scores indicating greater motor dysfunction. The total score for Part III ranges from 0 to 132, which is the sum of the individual item scores.
  The sum of the MDS-UPDRS Part II and Part III total scores ranges from 0 to 184, with high scores indicating greater clinical impairment.
Time Frame: Part 1: Week 40 and Part 2: Week 76
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- K0706, Low Dose: K0706: low dose, orally, once-daily in Parts 1 and 2
- K0706, High Dose: K0706: high dose, orally, once-daily in Parts 1 and 2 (in addition, participants who received placebo in Part 1 were transitioned to K0706, high dose in Part 2)
- Placebo: placebo: placebo, orally, once-daily (participants who received placebo in Part 1 were transitioned to K0706, high dose in Part 2)
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
score on a scale
  Part 1 Period: MDS-UPDRS (Sum of Parts II and III Total Scores) | 2.6 (10.83) | 2.7 (9.72) | -0.6 (9.53)
  Part 2 Period: MDS-UPDRS Part III Tremors Subscore: number analyzed (Participants) | 70 | 35 | 71
  Part 2 Period: MDS-UPDRS Part III Tremors Subscore | 0.4 (1.87) | -0.9 (2.54) | -0.4 (2.68)
  Part 2 Period: MDS-UPDRS Part III Bradykinesia Subscore: number analyzed (Participants) | 70 | 35 | 71
  Part 2 Period: MDS-UPDRS Part III Bradykinesia Subscore | -0.7 (2.25) | -0.1 (0.83) | 0.0 (2.20)
  Part 2 Period: MDS-UPDRS Part III Rigidity Subscore: number analyzed (Participants) | 70 | 35 | 71
  Part 2 Period: MDS-UPDRS Part III Rigidity Subscore | 1.7 (4.46) | 0.2 (3.81) | 0.8 (4.12)
  Part 2 Period: MDS-UPDRS Part III Axial Symptoms Subscore: number analyzed (Participants) | 70 | 35 | 71
  Part 2 Period: MDS-UPDRS Part III Axial Symptoms Subscore | 0.5 (1.22) | 0.4 (1.15) | 0.0 (1.37)

4. Secondary Outcome: To Determine if K0706 Delays the Initiation of Symptomatic Medications in Participants
Time Frame: Part 1: Week 40 and Part 2: Week 80 (Part 2 is applicable to the subjects who complete the EoT visit of part 1 (V11/Week 40) and who confirm their willingness to participate in part 2 of the study.
Population: Efficacy analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: placebo: placebo, orally, once-daily This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. Subjects that had been randomized to either dose of K0706 in part 1 of the study will continue on the same dosing regimen in Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
Participants | 149 | 129 | 144

5. Secondary Outcome: Change in Health Related Quality of Life as Measured by the European Quality of Life Questionnaire 5 Level Version
Description: Health-Related quality of life (HRQoL) will be measured using the European Quality of Life Questionnaire 5 level version (EQ-5D-5L). This scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.
Time Frame: Week 40
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
score on a scale | -0.0419 (0.11060) | -0.0531 (0.16289) | -0.0140 (0.10787)

6. Secondary Outcome: Change in Clinician Global Impression Severity
Description: The Clinician Global Impression Severity (CGIS) is a tool used to measure overall disease severity, assessed as follows:
  1. Normal
  2. Borderline
  3. Mild
  4. Moderate
  5. Marked
  6. Severe
  7. Among the Most Extremely Ill Patient
Time Frame: Week 40
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
score on a scale | 0.2 (0.68) | 0.0 (0.74) | 0.2 (0.91)

7. Secondary Outcome: Change in the Scales for Outcomes in Parkinson's Disease - Autonomic Questionnaire
Description: The Scales for Outcome in Parkinson's disease - Autonomic (SCOPA-AUT) sum score is a sum of rating scores over 23 items. The SCOPA-AUT sum score ranges from 0 to 69. A higher score means a more severe autonomic dysfunction (i.e., a worse outcome). For each of the 23 items, the score ranges from 0 to 3. The rating scale is the follows:
  0= Never experiencing the symptom;
  1. Sometimes experiencing the symptom;
  2. Regularly experiencing the symptom;
  3. Often experiencing the symptom
Time Frame: Week 40
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- K0706, Low Dose: K0706: low dose, orally, once-daily. This study consists of two parts. Subjects who had been randomized to placebo in Part 1 will be rolled over to a high dose K0706 (384 mg powder for suspension or equivalent formulation) at Week 40. Subjects that had been randomized to either dose of K0706 in part 1 of the study will continue on the same dosing regimen in Part 2 of the study. All subjects will continue treatment for up to 36 weeks.
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 164 | 162 | 161
score on a scale | 1.6 (7.70) | 3.8 (10.11) | 0.3 (7.76)

8. Secondary Outcome: Serum Concentration Level of K0706
Description: Plasma pharmacokinetic (PK) samples were collected Week 28, per the Schedule of Assessment of the study protocol. There was no PK samples collected after Week 28 per the study protocol.
Time Frame: Week 28
Population: PK Analysis Set (Part 1): The PK Analysis Set (Part 1) included all subjects who received at least one dose of study drug in Part 1 (i.e., the 40-week double-blind part) of the study and also had at least one blood sample taken to measure the K0706 concentration level.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | K0706, Low Dose | K0706, High Dose | Placebo
Number analyzed (Participants) | 151 | 150 | 0
ng/mL | 1127.8 (1379.69) | 1451.9 (1371.79) |

9. Other Pre Specified Outcome: Exploratory Outcome: Effect of K0706 on Dopamine Cell Health in Parkinson's Disease as Detected Via Dopamine Transporter Single Photon Emission Computed Tomography (DaT SPECT) Brain Imaging
Description: Not available: The results of the exploratory analyses, including examination of CSF using the α-synuclein aggregation assay and measurement of neurofilament light, were not intended for interpretation of efficacy.
Time Frame: Week 40
Reporting Status: Not Posted

10. Other Pre Specified Outcome: CSF K0706 Levels Progression or Target Engagement of K0706.
Description: as for outcome 9
Time Frame: Week 40
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Brain DaT SPECT - an Imaging Tool That is a Marker of Dopaminergic Cell Health.
Description: as for outcome 9
Time Frame: Week 40
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Blood K0706 Levels
Description: as for outcome 9
Time Frame: Week 40
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Skin Punch Biopsy
Description: as for outcome 9
Time Frame: Week 40
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Any AE/SAE that occurs until the follow-up visit, 30 days post Week 76 (the end of treatment visit), or 30 days post the last dose of study drug for subjects with early discontinuation, should be reported and included in the safety analysis of the study. Any AE/SAE occurring past this date will be reported only if it is considered related to study drug by the Investigator.
Description: Part 2 is an optional long-term extension study; patients who had previously received placebo were transitioned to high-dose K0706 in the part 2 study.
Groups:
- K0706, Low Dose (Part 2); K0706, Low Dose (Part 1): K0706: low dose, orally, once-daily
- K0706, High Dose (Part 2); K0706, High Dose (Part 1): K0706: high dose, orally, once-daily
- Placebo (Part 2): Prior placebo transitioned to K0706 high dose
- Placebo (Part 1): placebo: placebo, orally, once-daily
Arm/Group | K0706, Low Dose (Part 2) | K0706, High Dose (Part 2) | Placebo (Part 2) | K0706, Low Dose (Part 1) | K0706, High Dose (Part 1) | Placebo (Part 1)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/117 | 0/0 | 1/171 | 0/173 | 0/167
Serious Adverse Events (participants affected / at risk) | 3/72 | 11/117 | 0/0 | 14/171 | 7/173 | 5/167
Other Adverse Events (participants affected / at risk) | 21/72 | 85/117 | 0/0 | 131/171 | 150/173 | 124/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K0706, Low Dose (Part 2) (N=72) | K0706, High Dose (Part 2) (N=117) | Placebo (Part 2) (N=0) | K0706, Low Dose (Part 1) (N=171) | K0706, High Dose (Part 1) (N=173) | Placebo (Part 1) (N=167)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 2 (2)
Coronary Heart Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K0706, Low Dose (Part 2) (N=72) | K0706, High Dose (Part 2) (N=117) | Placebo (Part 2) (N=0) | K0706, Low Dose (Part 1) (N=171) | K0706, High Dose (Part 1) (N=173) | Placebo (Part 1) (N=167)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (9) | 0 (0) | 9 (10) | 16 (20) | 13 (17)
Nasopharyngitis (Infections and infestations) | 4 (6) | 3 (3) | 0 (0) | 5 (7) | 6 (7) | 12 (13)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 11 (13) | 13 (15) | 10 (12)
Tremor (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 6 (6) | 14 (14) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 18 (22) | 18 (22) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 0 (0) | 18 (18) | 20 (30) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (10) | 0 (0) | 23 (28) | 30 (34) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9) | 0 (0) | 9 (13) | 18 (19) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 10 (11) | 14 (17) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 6 (6) | 0 (0) | 14 (16) | 5 (7) | 9 (9)
Fatigue (General disorders) | 0 (0) | 8 (8) | 0 (0) | 5 (11) | 17 (20) | 8 (8)
Covid-19 (Infections and infestations) | 0 (0) | 6 (6) | 0 (0) | 17 (17) | 7 (7) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 10 (10) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 5 (8) | 9 (9) | 6 (7)
Dizziness (Nervous system disorders) | 2 (3) | 3 (5) | 0 (0) | 4 (4) | 10 (12) | 8 (12)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 10 (12) | 8 (8)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 7 (7) | 12 (14) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 5 (6) | 8 (11) | 2 (4)
Asthenia (General disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03655236/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03655236/SAP_001.pdf